CLINICAL TRIAL: NCT00886873
Title: Mifepristone 5 mg Versus 10 mg During 6 Months for the Treatment of Uterine Leiomyomata. A Randomized, Double Blinded Clinical Trial.
Brief Title: Mifepristone 10 or 5 mg for 6 Months to Treat Uterine Fibroids
Acronym: Mifemyo_2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mediterranea Medica S. L. (Other)
Responsible Party: Principal Investigator, Dr. Josep Lluis Carbonell i Esteve, Medical Director, Mediterranea Medica S. L.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mife_Fibroids_02
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; Mifepristone; Antiprogestins
MeSH Terms: conditions — Leiomyoma | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Oral administration of mifepristone 5 mg daily for six months.
  Interventions: Drug: Mifepristone
- Group 2 (Experimental): Oral administration of mifepristone 10 mg daily for six months.
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
The objectives of this study are to estimate the efficacy and safety of the daily administration for 6 months of 5 mg versus 10 mg. A 6 month follow-up of subjects is carried out to estimate how the effects of mifepristone are kept in time.

The hypothesis of this study is that both mifepristone doses reduce the volume of the myoma up to 50% in six months treatment.

DETAILED DESCRIPTION:
Women, in fertile age or premenopausal status, presenting symptomatic myomaswere randomly assigned to receive 5 or 10 mg of mifepristone for six months.

The decreasing in the prevalence of symptoms attributable to myomas is an important goal to achieve under both treatments. Another goal is to maintain for more than 6 months the benefits of the treatment with mifepristone.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine fibroids
* Reproductive age or premenopausal
* Accepting the use of non hormonal contraception
* Conformity in keeping a monthly log of all episodes of vaginal bleeding during the treatment as well as the side effects of mifepristone
* Agreeing to have ultrasound examinations in every follow-up or evaluation visit
* Agreeing in two endometrial biopsies: one before starting treatment and another in the following 10 days after treatment termination

Exclusion Criteria:

* Pregnancy or desire to become pregnant
* Breastfeeding
* Hormonal contraception or any hormonal therapy received in the last three months
* Signs or symptoms of pelvic inflammatory disease
* Adnexal masses
* Abnormal or unexplained vaginal bleeding
* Suspected or diagnosed malignant neoplastic disease
* Signs or symptoms of mental illness
* Adrenal disease
* Sickle cell anemia
* Hepatic disease
* Renal disease
* Coagulopathy
* Any other severe or important disease
* Any contraindication to receiving antiprogestins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Volume of the uterine leiomyomata with 5 versus 10 mg of mifepristone daily after six months of treatment | 6 months

SECONDARY OUTCOMES:
Prevalence of symptoms after 6 months treatment with 5 or 10 mg of mifepristone. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carbonell Josep Ll., MD, Principal Investigator — Mediterranea Medica S. L.
Locations (1):
- Hospital Eusebio Hernandez, Ciudad Habana, La Habana, Cuba